CLINICAL TRIAL: NCT05322876
Title: Feasibility of Reducing Cardiovascular Disease Risk Factors in Hispanics Through a Family-Based Community Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Poudre Valley Health System (Other)
Collaborators: Fitbit LLC (Industry)
Responsible Party: Principal Investigator, Gary J. Luckasen, MD, Principal Investigator, Poudre Valley Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HHFP-001
Record Dates: First submitted 2022-02-25; First posted 2022-04-12 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Cardiovascular Diseases; Metabolic Syndrome
Keywords: Metabolic Syndrome; Cardiovascular Disease Risk Factors; Community Intervention
MeSH Terms: conditions — Cardiovascular Diseases; Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: Sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy Hearts Family Program (Experimental): Participants will be enrolled in the standard Healthy Hearts Family Program 6-month family-based cardiovascular disease prevention program.
  Interventions: Behavioral: Healthy Hearts Family Program

INTERVENTIONS:
Behavioral: Healthy Hearts Family Program — Participants will participate in a baseline health and knowledge screening, followed by a 6-week once-weekly class series, and 3- and 6-month follow-up health and knowledge screenings.

SUMMARY:
The purpose of this study is to evaluate the feasibility of a 6-month family-based community intervention to mitigate cardiovascular disease risk factors in Hispanic families in northern Colorado as measured through biometric screenings, body composition, physical activity, and health knowledge.

DETAILED DESCRIPTION:
The current project aims to leverage the UCHealth Healthy Hearts Family Program to provide a free, non-insurance-based 1-year cardiovascular disease (CVD) prevention and wellness program to Hispanic Colorado families. This program includes an interactive educational class series, baseline and quarterly biometric screenings, and optional consultations with an Exercise Physiologist and a Dietitian. This program takes a novel approach to preventative care by incorporating the family unit with the intention of having the child be the agent of change. The long-term goals of this project are to significantly improve CVD risk factors among participating families and to disseminate study findings to inform developing and current outreach programs to offer effective CVD prevention programs for Hispanic citizens. This work may ultimately lead to more Hispanics being served through new or existing programs, therefore expanding important preventative community health interventions into this underserved population.

ELIGIBILITY:
Inclusion Criteria:

* At least one member of the family unit self-identifies as Hispanic
* At least 13 years of age

Exclusion Criteria:

* Unwilling to wear Fitbit devices daily for 6 months except when charging and sleeping
* Cannot read or understand either English or Spanish
* Cannot return to screening location to perform the minimum of the baseline, 3-month and 6-month follow-up screenings
* Children or adolescents will be excluded from this project without a minimum of one accompanying parent or guardian

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-03-22 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy of program through changes in physical health - Daily Steps | Baseline, 3-month follow up and 6-month follow up data will be evaluated and compared
  Physical activity metrics (daily average steps per month) measured by Fitbit devices
Efficacy of program through changes in physical health - Physical Activity | Baseline, 3-month follow up and 6-month follow up data will be evaluated and compared
  Physical activity metrics (daily minutes of light, moderate and vigorous activity per month) measured by Fitbit devices
Efficacy of program through changes in physical health - Blood Pressure | Baseline, 3-month follow up and 6-month follow up data will be evaluated and compared
  Biometric variables (blood pressure in mmHg)
Efficacy of program through changes in physical health - Lab Value -Lipid Profile | Baseline, 3-month follow up and 6-month follow up data will be evaluated and compared
  Biometric variables - lab values (lipid profile in mg/dL) measured through finger stick blood sampling
Efficacy of program through changes in physical health - Lab Value - Triglycerides | Baseline, 3-month follow up and 6-month follow up data will be evaluated and compared
  Biometric variables - lab values ( triglycerides in mg/dL) measured through finger stick blood sampling
Efficacy of program through changes in physical health - Lab Value - Blood Glucose | Baseline, 3-month follow up and 6-month follow up data will be evaluated and compared
  Biometric variables - lab values (blood glucose all in mg/dL) measured through finger stick blood sampling
Efficacy of program through changes in physical health - Waist Circumference | Baseline, 3-month follow up and 6-month follow up data will be evaluated and compared
  Body composition (waist circumference in inches)
Efficacy of program through changes in physical health - Body Composition - Muscle Mass | Baseline, 3-month follow up and 6-month follow up data will be evaluated and compared
  Body composition (muscle mass in pounds) measured with a Tanita MC980Uplus multi-frequency bio-electrical impedance analysis device.
Efficacy of program through changes in physical health - Body Composition - Fat Mass | Baseline, 3-month follow up and 6-month follow up data will be evaluated and compared
  Body composition (fat-free mass in pounds) measured with a Tanita MC980Uplus multi-frequency bio-electrical impedance analysis device.
Efficacy of program through changes in physical health - Body Fat Percentage | Baseline, 3-month follow up and 6-month follow up data will be evaluated and compared
  Body composition (body fat percentage) measured with a Tanita MC980Uplus multi-frequency bio-electrical impedance analysis device.
Efficacy of program through changes in physical health - Visceral Fat Rating | Baseline, 3-month follow up and 6-month follow up data will be evaluated and compared
  Body composition (Tanita visceral fat rating) measured with a Tanita MC980Uplus multi-frequency bio-electrical impedance analysis device.
Efficacy of program through changes in health knowledge | Baseline, post-6 week class series, 3- and 6-month follow-up appointments.
  Health knowledge gained and retained will be evaluated and compared at baseline, post-6 week class series, 3- and 6-month follow-ups utilizing previously developed and utilized Healthy Hearts knowledge survey. This outcome will be measured by correct responses on the Healthy Hearts knowledge survey.

SECONDARY OUTCOMES:
Adherence to program and utilization of additional resources - Program attendance - Percentage of Scheduled Visits Attended | These variables will be measured and assessed throughout the full 6 month program.
  Attendance for screenings, classes and other consultations across baseline and follow-up visits. Attendance will be measured as the percentage of scheduled visits (including the 6 week class series and the 3- and 6-month follow-up visits) completed.
Adherence to program and utilization of additional resources - Fitbit Utilization | These variables will be measured and assessed throughout the full 6 month program.
  Compliance to Fitbit utilization as measured by days worn throughout the 6 month program. The NHANES compliance to wear time of > 10 hours worn per day will be utilized.
Adherence to program and utilization of additional resources - Resource Utilization | These variables will be measured and assessed throughout the full 6 month program.
  Use of Exercise Physiologist and Dietician resources provided will be quantified and reported. This outcome will be reported as the number of consultation appointments requested and utilized throughout the program.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Bandera, MS, Principal Investigator — University of Colorado Health
Locations (1):
- Medical Center of the Rockies, Loveland, Colorado, United States

IPD SHARING:
Plan to Share IPD: No